CLINICAL TRIAL: NCT01249261
Title: A 1-year, Risedronate-free, Multicenter, Outpatient, Phase IIIb Extension Study to Assess Bone Turnover Recovery in Women With Postmenopausal Osteoporosis Who Sequentially Completed Clinical Studies RVE009093, RVE1996077, and RVE1998080 (no NCT Study Numbers)
Brief Title: Effect of Stopping Risedronate After Long Term Treatment on Bone Turnover
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001079
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Postmenopausal Women With Osteoporosis
Keywords: Postmenopausal Women; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo/Risedronate (Placebo Comparator): Placebo years 1-5, Risedronate 5mg/day years 6 & 7, no drug year 8
  Interventions: Drug: Placebo/Risedronate
- Risedronate (Active Comparator): Risedronate 5mg years 1-7, no drug year 8
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — 5 mg/day
  Arms: Risedronate
Drug: Placebo/Risedronate — placebo years 1-5 followed by 5 mg risedronate years 6 & 7 and no drug year 8
  Arms: Placebo/Risedronate

SUMMARY:
The effects of stopping long-term (7 years) and short term (2 years) risedronate therapy on BMD (bone mineral density) and BTMs (bone turnover markers) will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women who sequentially completed studies RVE009093, RVE1996077, RVE1998080

Exclusion Criteria:

* Less than 60% compliant between drug start and month 21
* Using bisphosphonates, glucocorticoids, anabolic steroids, vitamin D supplements, calcitrol, estrogen or estrogen-related drugs, progestogen, depot injection >10,000 IU vitamin D, investigational drug

Max Age: 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2001-10; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (10):
- Australia (2):
  - Investigational Site, Concord, New South Wales
  - Investigational Site, Parkville, Victoria
- Investigational Site, De Pintelaan 185, Gent, Belgium
- Investigational Site, Hvidovre, Denmark, Denmark
- Investigational Site, Oulu, Finland, Finland
- Investigational Site, Siena, Italy, Italy
- Investigational Site, Warsaw, Poland, Poland
- Spain (2):
  - Investigational Site, Barcelona, Spain
  - Investigational Site, Madrid, Spain
- Investigational Site, Gothenburg, Sweden, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began 4 October 2001
Pre-assignment Details: Patients who sequentially completed Clinical Studies RVE009093 (3 year core study), RVE1996077 Year 4/5 extension study) and RVE1998080 (Year 6/7 extension study) were eligible for screening. [No NCT numbers available]
Period: Overall Study
Arm/Group | Placebo/Risedronate | Risedronate
Started | 30 | 31
Completed | 29 | 31
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Risedronate | Risedronate | Total
Number analyzed (Participants) | 30 | 31 | 61
Age Continuous [Mean (Standard Deviation); unit: Participants] | 66.9 (6.24) | 67.3 (5.79) | 67.1 (5.97)
Age, Customized [Number; unit: Participants]
  < 65 years old | 11 | 9 | 20
  > or = 65 years old | 19 | 22 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  Finland | 1 | 3 | 4
  Spain | 5 | 7 | 12
  Poland | 8 | 9 | 17
  Belgium | 0 | 2 | 2
  Denmark | 5 | 3 | 8
  Australia | 4 | 3 | 7
  Italy | 3 | 1 | 4
  Sweden | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Lumbar Spine Bone Mineral Density (BMD) From Core Study Baseline, Month 6, Intention to Treat (ITT) Population
Description: Hologic or Lunar Machines: same equipment used in prior study should be used for all patient visits. sBMD (standardized BMD): Lunar sBMD = 952.2*BMD, Hologic sBMD = 1075.5*BMD. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 6 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | 6.2217 (1.82459) | 12.7784 (2.09663)

2. Primary Outcome: Mean Percent Change in Lumbar Spine BMD From Core Study Baseline, Month 12, ITT Population
Description: as for outcome 1
Time Frame: Baseline Core Study (Year 1) to Month 12 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | 5.5312 (1.66394) | 13.3472 (2.09761)

3. Primary Outcome: Mean Percent Change in Lumbar Spine BMD From Core Study Baseline, Month 12/Endpoint, ITT Population
Description: Endpoint is the last measurement during the 12 month treatment period during Year 8. Hologic or Lunar Machines: same equipment used in prior study should be used for all patient visits. sBMD (standardized BMD): Lunar sBMD = 952.2*BMD, Hologic sBMD = 1075.5*BMD. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 12/Endpoint (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | 5.5312 (1.66394) | 13.3472 (2.09761)

4. Primary Outcome: Mean Percent Change in Femoral Neck BMD From Core Study Baseline, Month 6, ITT Population
Description: Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. Normalized baseline femoral neck BMD lunar equipment only 0.836*BMD - 0.008; Hologic reference. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 6 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | -1.0384 (2.19722) | 1.4797 (1.03811)

5. Primary Outcome: Mean Percent Change in Femoral Neck BMD From Core Study Baseline, Month 12, ITT Population
Description: as for outcome 4
Time Frame: Baseline Core Study (Year 1) to Month 12 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | -0.2530 (1.83321) | 3.2192 (3.55882)

6. Primary Outcome: Mean Percent Change in Femoral Neck BMD From Core Study Baseline, Month 12/Endpoint, ITT Population
Description: Endpoint is the last measurement during the treatment period (thru Month 12, Year 8). Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. Normalized baseline femoral neck BMD lunar equipment only 0.836*BMD - 0.008; Hologic reference. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 12/Endpoint (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | -1.1148 (1.94506) | 3.2192 (3.55882)

7. Primary Outcome: Mean Percent Change in Femoral Trochanter BMD From Core Study Baseline, Month 6, ITT Population
Description: Month 6, Year 8 compared to Baseline, Year 1. Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 6 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | 1.6386 (1.39295) | 4.4060 (1.54420)

8. Primary Outcome: Mean Percent Change in Femoral Trochanter BMD From Core Study Baseline, Month 12, ITT Population
Description: Baseline, year 1 compared with Month 12, year 8. Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 12 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | 1.9561 (1.37883) | 2.2334 (1.37500)

9. Primary Outcome: Mean Percent Change in Femoral Trochanter BMD From Core Study Baseline, Month 12/Endpoint, ITT Population
Description: Endpoint is the last measurement during the treatment period (through Month 12, Year 8) compared with baseline Year 1. Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 12/Endpoint (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | 1.4058 (1.42232) | 2.2334 (1.37500)

10. Primary Outcome: Mean Percent Change in Total Proximal Femur BMD From Core Study Baseline, Month 6, ITT Population
Description: Baseline, Year 1 compared with Month 6, Year 8. Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 6 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | -1.3867 (1.98837) | 3.3871 (0.96971)

11. Primary Outcome: Mean Percent Change in Total Proximal Femur BMD From Core Study Baseline, Month 12, ITT Population
Description: as for outcome 8
Time Frame: Baseline Core Study (Year 1) to Month 12 (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | -2.2999 (1.67680) | 0.6672 (0.99708)

12. Primary Outcome: Mean Percent Change in Total Proximal Femur BMD From Core Study Baseline, Month 12/Endpoint, ITT Population
Description: Baseline, Year 1 compared with Endpoint (last measurement during the treatment period through Month 12), Year 8. Allowed equipment Hologic or Lunar. Same equipment used in prior study should be used for all patient visits. All scans analyzed centrally by Synarc (Portland, OR).
Time Frame: Baseline Core Study (Year 1) to Month 12/Endpoint (Year 8)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo/Risedronate | Risedronate
Number analyzed (Participants) | 30 | 31
Percent Change | -3.2799 (1.80579) | 0.6672 (0.99708)

ADVERSE EVENTS:
Time Frame: Twelve months treatment free period.
Arm/Group | Placebo/Risedronate | Risedronate
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/31
Other Adverse Events (participants affected / at risk) | 18/30 | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Risedronate (N=30) | Risedronate (N=31)
Accidental Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Risedronate (N=30) | Risedronate (N=31)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (4) | 1 (1)
Accidental Injury (Injury, poisoning and procedural complications) | 3 (5) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Neurosis (Nervous system disorders) | 0 (0) | 1 (1)
Sleep Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
ExtraPyramidal Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hyperkinesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1)
Peripheral Vascular Disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Traumatic Bone Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermatologic Fungus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Amblyopia (Eye disorders) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased GGTP (Gamma Glutamyl Transpeptidase) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (3) | 1 (2)
Endometrial Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less